CLINICAL TRIAL: NCT00705081
Title: Observational Study Evaluating the LDL-C Lowering Effects of Ezetimibe With a Statin as Prescribed in Daily Routine Practice in an Indonesian Population
Brief Title: Evaluation of the LDL-C Lowering Effects of Ezetimibe Achieved in Co-administration Therapy With Statins in an Indonesian Population (Study P04276)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P04276
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Not previously treated: subjects with hypercholesterolemia, who had never been treated with any cholesterol-lowering agent, and received the combination of ezetimibe 10 mg and a statin as initiation therapy
  Interventions: Drug: ezetimibe; Drug: statin
- Previously treated with statin: subjects with hypercholesterolemia, who were previously treated with a statin, and received ezetimibe 10 mg as add-on therapy
  Interventions: Drug: ezetimibe; Drug: statin

INTERVENTIONS:
Drug: ezetimibe — 10 mg once daily
  Other Names: SCH 58235
Drug: statin

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the low-density lipoprotein-cholesterol (LDL-C) lowering in an Indonesian population treated with ezetimibe co-administered with a statin in routine daily practice. In addition, the study will investigate whether and to what extent the target levels set by the participating doctors are achieved by the co-administration therapy.

DETAILED DESCRIPTION:
Sampling method: invitation to the physician's patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects that were to receive ezetimibe 10 mg as prescribed in daily practice

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects with hypercholesterolemia
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Not Previously Treated | Previously Treated With Statin
Started | 255 | 198
Completed | 255 | 198
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Previously Treated | Previously Treated With Statin | Total
Number analyzed (Participants) | 255 | 198 | 453
Age, Customized [Number; unit: participants]
  20-30 years | 4 | 1 | 5
  31-40 years | 21 | 9 | 30
  41-50 years | 69 | 57 | 126
  51-60 years | 108 | 81 | 189
  >61 years | 53 | 50 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 79 | 185
  Male | 149 | 119 | 268
Region of Enrollment [Number; unit: participants]
  Indonesia | 255 | 198 | 453

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events
Description: Safety and tolerability of LDL lowering with co-administration therapy as measured by the number of participants reporting adverse events (AE). (AE defined as any untoward medical occurrence or unfavorable and unintended sign in a subject administered the pharmaceutical product whether or not considered related to the use of that product.)
Time Frame: 4-6 weeks after the first visit
Population: All participants enrolled
Measure: Number; unit: Participants
Arm/Group | Not Previously Treated | Previously Treated With Statin
Number analyzed (Participants) | 255 | 198
Participants | 1 | 1

2. Primary Outcome: Intensity of Adverse Events Reported
Description: Intensity of adverse events reported after co-administration therapy
Time Frame: 4-6 weeks after the first visit
Population: All participants enrolled
Measure: Number; unit: Participants
Arm/Group | Not Previously Treated | Previously Treated With Statin
Number analyzed (Participants) | 255 | 198
Participants
  Mild | 1 | 1
  Moderate | 0 | 0
  Severe | 0 | 0

3. Primary Outcome: Participants Achieving Low-density Lipoprotein-cholesterol (LDL-C) Target Levels With Co-administration Therapy
Description: Achievement of LDL-C target levels as determined by physician
Time Frame: 4-6 weeks after the first visit
Population: All patients enrolled
Measure: Number; unit: Participants
Arm/Group | Not Previously Treated | Previously Treated With Statin
Number analyzed (Participants) | 255 | 198
Participants | 101 | 106

ADVERSE EVENTS:
Arm/Group | Not Previously Treated | Previously Treated With Statin
Serious Adverse Events (participants affected / at risk) | 0/255 | 0/198
Other Adverse Events (participants affected / at risk) | 0/255 | 0/198

LIMITATIONS AND CAVEATS:
Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less